CLINICAL TRIAL: NCT06080035
Title: Open-label, Prospective Study on the Effects of Cetyl Tranexamate Mesylate on the Appearance of Acne-Related Hyperpigmentation
Brief Title: The Effects of Cetyl Tranexamate Mesylate on the Appearance of Acne-Related Hyperpigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Actera (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i23-01_CTM
Record Dates: First submitted 2023-10-02; First posted 2023-10-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hyperpigmentation; Post-inflammatory Hyperpigmentation; Acne
MeSH Terms: conditions — Hyperpigmentation; Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical Cetyl Tranexamate Mesylate (Experimental): Product will be used on the face twice daily in the morning and in the evening for 2 weeks.
  Interventions: Other: Topical Cetyl Tranexamate Mesylate

INTERVENTIONS:
Other: Topical Cetyl Tranexamate Mesylate — Topical product will be applied onto clean skin morning and night.

SUMMARY:
The purpose of this study is to assess the effects of Cetyl Tranexamate Mesylate on acne-related hyperpigmentation through a specific delivery form known as TeraCeutic TXVector.

DETAILED DESCRIPTION:
Hyperpigmentation is characterized as an increase in pigment on the skin and is a common skin condition in individuals with skin types III to VI on the Fitzpatrick skin classification scale. Hyperpigmentation can be localized to an area in the form of post-inflammatory hyperpigmentation or diffused in the form of melasma. One of the treatments that are used to treat hyperpigmentation is tranexamic acid (TXA) which is a third-generation bioactive and is formally known to work as a plasmin inhibitor. Since TXA is hydrophilic in nature and has a strong hydrogen-bonding capacity, it has an insufficient skin permeability. Similar to TXA esters, Cetyl Tranexamate Mesylate (CTM) is hypothesized to have greater permeability and this study will evaluate the effects of CTM on the appearance of post-inflammatory hyperpigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 14 years of age until 55 years of age
* Individuals experiencing 3 different areas minimum of facial post-inflammatory hyperpigmentation in those with acne

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners.
* Adults unable to consent.
* Those who are unwilling to discontinue hydroquinone, vitamin A/C/E, azelaic acid, kojic acid, bakuchiol, licorice root, retinol, niacinamide, alpha arbutin, and oral or topical tranexamic acid for two weeks to meet the washout criteria prior to enrolling and for the duration of the study.
* Subjects with any of the following facial cosmetic treatments within the past 3 months or those who are unwilling to withhold the following facial cosmetic treatments during study including microdermabrasion, intense pulsed light (IPL), peels, laser treatments, acid treatments, or any other medical treatment administered by a physician or skin care professional which is designed to improve skin pigmentation.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Facial skin pigment intensity of 3 pre-identified lesions | 2 weeks
  Change in the appearance of pigment intensity (melanin measurement) of 3 pre-identified hyperpigmented lesions

SECONDARY OUTCOMES:
Facial skin pigment intensity of 3 pre-identified lesions | 1 week
  Change in the appearance of pigment intensity (melanin measurement) of 3 pre-identified hyperpigmented lesions
Self-perception of skin pigmentation | 1 week
  Survey-based self-assessment of facial skin pigmentation
Self-perception of skin pigmentation | 2 week
  Survey-based self-assessment of facial skin pigmentation
Self-perception of skin redness | 1 week
  Survey-based self-assessment of aspects of skin redness
Self-perception of skin redness | 2 week
  Survey-based self-assessment of aspects of skin redness

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD MS AP, Principal Investigator — Integrative Skin Science and Research
Locations (1):
- Integrative Skin and Research, Sacramento, California, United States